CLINICAL TRIAL: NCT04769440
Title: Effect of MgSo4 Infusion on Oxygenation and Lung Mechanics in Morbidly Obese Patients Undergoing Bariatric Surgery.A Randomized Clinical Trial
Brief Title: Effect of mgso4 on Oxygenation and Lung Mechanics in Morbidly Obese Patients During Bariatric Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Marwa Mostafa Mohamed Ali Mowafi, Lecturer of anesthesia ,principal Investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FMASU R 07/2021
Record Dates: First submitted 2021-02-14; First posted 2021-02-24 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Anesthesia
Keywords: mgso4; oxygenation; lung mechanics
MeSH Terms: interventions — Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- M group (Mg sulphate ) (Active Comparator): patients will receive 30mg/kg LBW of 10%mgso4 in 100 ml normal saline intravenously over 30 minutes as a loading dose ,followed by 10 mg /kg LBW for 90 minutes
  Interventions: Drug: mg sulphate
- C group (control ) (No Intervention): patients will receive 100 ml of normal saline intravenously over 30 minutes followed by saline infusion for 90 minutes

INTERVENTIONS:
Drug: mg sulphate — mgso4 infusion will start 15 minutes after intubation , 30 mg/kg LBW of 10%mgso4 in 100 ml normal saline I.V ,over 30 minutes followed by 10 mg/kg LBW for 90 minutes
  Other Names: mgso4
  Arms: M group (Mg sulphate )

SUMMARY:
The purpose of this trial is to study the effect of mgso4 infusion on oxygenation and lung mechanics in morbidly obese patients undergoing bariatric surgery

DETAILED DESCRIPTION:
Background and objectives: morbidly obese patients are characterized by a high prevalence of restrictive lung disease. Respiratory mechanics are significantly altered in obesity. These changes are exacerbated with general anesthesia .Obesity also results in reduced lung and chest wall compliance ,increased lung resistance ,reduced oxygenation.MgSo4 is promising in managing several respiratory disorders.it cause smooth muscle relaxation and reduce airflow obstruction.

The objective of this trial is to study the effect of mgso4 infusion on oxygenation and lung mechanics in morbidly obese patients undergoing bariatric surgery.

the following will be recorded :intraoperative oxygenation,lung mechanics,MAP,HR,EtCO2,plateau and peak airway pressure,sedation score,serum mgso4 level,change in P/F ratio and dynamic lung compliance,respiratory rate postoperative

ELIGIBILITY:
Inclusion Criteria:

* Patients age between 21-60 years.
* BMI more than 40kg/m2
* Patients with restrictive lung disease(FVC>70%)
* American society of Anesthesiologists(ASA) physical status II
* No previous abdominal surgery
* Scheduled for laparoscopic bariatric surgery not exceeding 3 hours.

Exclusion Criteria:

* Patient refusal to participate in the study
* ASA physical status more than II
* patients with heart failure
* Kidney disease
* Patients on antiarrhythmic drugs
* Patients taking beta or calcium channel blockers
* Allergy to study drugs
* Patients with combined restrictive-obstructive lung disease

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-02-03 (Actual); Study Completion 2022-02-21 (Actual)

PRIMARY OUTCOMES:
Pao2 | 5 minutes after intubation to 90 minutes after starting drug infusion
  arterial oxygenation during surgery determined by Pao2
Pao2/FIO2 | 5 minutes after intubation to 90 minutes after starting drug infusion
  arterial oxygenation during surgery determined by Pao2/FIO2

SECONDARY OUTCOMES:
Static lung compliance | 5 minutes after intubation to 90 minutes after starting drug infusion
  will be calculated as:tidal volume/(plateau pressure-positive end expiratory pressure)
mg sulphate level | One hour postoperatively
  serum mgso4 level
dead space | 5 minutes after intubation to 90 minutes after starting drug infusion
  dead space will be calculated as : Vd/Vt
Dynamic lung compliance | 5 minutes after intubation to 90 minutes after starting drug infusion
  will be calculated as :tidal volume/(peak airway pressure-positive end expiratory pressure)

CONTACTS AND LOCATIONS:
Overall Officials: Marwa M Mowafi, MD, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University Hospital, Cairo, Abassia, Egypt

IPD SHARING:
Plan to Share IPD: No